CLINICAL TRIAL: NCT04478929
Title: Early Detection of Cancer in Cases of Barrett's Esophagus Using Robotic Endoscopy Image Analysis Through Deep Image Retrieval
Brief Title: Early Detection of Barrett's Esophagus Through Deep Image Retrieval
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Leigh Taylor (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor-Investigator, Leigh Taylor, Senior Research Officer, University of the West of England
Organization: University of the West of England (Other)
Other Study IDs: REDM0227_RP01
Record Dates: First submitted 2020-07-15; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- gastroscopy clinic patients: NBT gastroscopy clinic invited participants. Patients are already due to attend the clinic, and we are inviting them to share their gastroscopy data with our research study.
  Interventions: Diagnostic Test: Gastroscopy

INTERVENTIONS:
Diagnostic Test: Gastroscopy — Routine gastroscopy

SUMMARY:
Barrett's oesophagus is a condition in which the area between the oesophagus and stomach no longer closes, allowing acidic contents of the stomach to enter the oesophagus and damage the lining. The project aims to assist clinicians by offering informed biopsy process, in which the system presents the operator with clinical outcomes of patients with visually similar GI tracts. The project goal is to assess the use of artificial intelligence-based similarity detection systems to better inform biopsy placement, increasing the reliability of bi-yearly inspections.

DETAILED DESCRIPTION:
The project intention is to acquire secondary endoscopy captured data from clinicians to create a sufficient dataset to train a learning system to achieve the stated objective. The data required will feature footage (images/videos) from inside the oesophagus. The preferred data would contain associated diagnosis notes and description, however, data without diagnosis can still be used. All data can and will be anonymised, as personal information will not be useful in this work.

The data will be labelled by either researchers, or professional clinicians and prepared ready to feed into a chosen learning AI system. Through an iterative learning process, the chosen AI system will learn to discriminate between severity of Barrett's oesophagus and output optimal biopsy target.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Attending Southmead Hospital for on OGD
* Has capacity
* Initially any indication, later patients with known Barrett's oesophagus

Exclusion Criteria:

* Children (<18)
* Patients without capacity
* Urgent and emergency procedures
* Limited English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Attending NBT clinic for on OGD phase 1, then later attending NBT clinic due to suspected Barrett's.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
gastroscopy image data set | 12 months
  Images collected during routine gastroscopy with examination notes

CONTACTS AND LOCATIONS:
Locations (1):
- NBT, Southmead Hospital, Bristol, Avon, United Kingdom

IPD SHARING:
Plan to Share IPD: No